CLINICAL TRIAL: NCT04809649
Title: SUBA-Itraconazole Therapy for Coccidioidomycosis Refractory or Intolerant to Fluconazole
Acronym: SITRIS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor is not proceeding with study due to budget cuts as a result of COVID-19.
Sponsor: George R Thompson (Other)
Collaborators: Mayne Pharma International Pty Ltd (Industry)
Responsible Party: Sponsor-Investigator, George R Thompson, Associate Professor of Medicine, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1666482
Record Dates: First submitted 2021-03-01; First posted 2021-03-22 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Coccidioidomycosis; Valley Fever
MeSH Terms: conditions — Coccidioidomycosis | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SUBA-itraconazole (Experimental): Drug: SUBA-itraconazole Dosage Form: 65 mg capsules Dosage: 260 mg/day Frequency: 130 mg twice daily (BID) Duration: Up to 180 days
  Interventions: Drug: SUBA-itraconazole

INTERVENTIONS:
Drug: SUBA-itraconazole — Participant will receive treatment with SUBA-itraconazole
  Other Names: Tolsura

SUMMARY:
The purpose of this study is to determine how safe, effective, and well tolerated a new investigational antifungal drug, SUBA-itraconazole, is for patients who have been previously treated with fluconazole and have had either an insufficient response to treatment with fluconazole or a negative reaction to fluconazole preventing their further treatment with it.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label study involving subjects with proven or probable coccidioidomycosis refractory to fluconazole therapy following >40 days of treatment or subjects with proven or probable coccidioidomycosis who are intolerant to fluconazole.

The availability "Super Bioavailability" (SUBA) itraconazole 65 mg capsules with twice-daily dosing options with improved pharmacokinetics and lack of food or acidity requirements offers a substantial opportunity to improve the treatment of subjects with coccidioidomycosis.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects ≥ 18 years who have given written informed consent to participate
2. Subjects with a proven or probable coccidioidomycosis according to current European Organisation for Research and Treatment of Cancer/Mycoses Study Group (EORTC/MSG) criteria, including subjects who:

   * Are immunosuppressed, including as a result of HIV/AIDS
   * Have had a heart, lung or bone marrow transplant
   * Have had chemotherapy for cancer
   * Are otherwise not immunocompromised

   Note: central nervous system (CNS) infection is an exclusionary criteria
3. Refractory for ≥ 40 days, or intolerant to fluconazole treatment for coccidioidomycosis in the opinion of the investigator

   * Refractory disease defined as failure to obtain an adequate therapeutic response after ≥40 days of therapy:
   * Lack of improvement in signs, symptoms or imaging findings OR
   * Continued isolate of Coccidioides or histopathologic findings of • Coccidioides despite antifungal therapy
   * Rising Complement Fixation Titers
   * Progression of disease (requires worsening of attributable signs, symptoms or imaging, or a new site of infection
   * Intolerance defined as adverse events attributable to fluconazole therapy defined as organ toxicity of grade 3 or higher, nephrotoxicity (Creatinine twice the upper limit of normal), or idiosyncratic reactions therapy that in the opinion of the investigator may be relieved by a therapeutic change OR refusal of the patient to take further fluconazole
4. Subjects of childbearing potential should be non-pregnant and not breastfeeding (and not planning to become pregnant)

   * Postmenopausal for ≥1 year
   * Post-hysterectomy or bilateral oophorectomy
   * If of child-bearing potential have a negative pregnancy test at screening and using an acceptable effective method of birth control throughout course of study or remain abstinent for duration of study. Subjects with a partner of childbearing potential should agree to use appropriate contraception.

Exclusion Criteria:

1. Significant liver dysfunction as evidenced by total bilirubin > 1.5 × the upper limit of normal (ULN) range unless considered due to Gilbert syndrome, in which case > 3 × the ULN, and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels > 1.5 x the ULN.
2. Evidence of CNS infection.
3. Unable to take PO medications.
4. Documented intolerance, allergy or hypersensitivity to itraconazole.
5. Inability to comply with study treatment, study visits, and study procedures.
6. Known history or presence of congestive cardiac failure, fungal endocarditis, or other causes of ventricular dysfunction that may outweigh the benefit of itraconazole.
7. Subjects with active tuberculosis.
8. Concurrent use of drugs that effect SUBA™-itraconazole concentrations

   • Subjects who washout from prohibited medications can be included
9. Any known or suspected condition of the subject that may jeopardize adherence to the protocol requirements or impede the accurate measurement of efficacy.
10. Treatment with any investigational agent in the 30 days prior to study entry.
11. Subjects unlikely to survive 30 days based on the opinion of the investigator.
12. Subjects with body weight < 40 kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-15 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
1. The Proportion of Participants Who Achieve Clinical Improvement, in All Participants Who Took at Least One Dose of Study Drug | 180 days
  Clinical Improvement is defined as at a) at least a 50% reduction in coccidioidomycosis Mycoses Study Group (MSG Score) from baseline value, or b) the unequivocal documentation of clinical improvement as recorded on the progress note of the medical provider, or c) a 25%-49% decrease in the MSG score from baseline value and a physician's impression of improvement as recorded on the progress note. The MSG score is a composite scoring system that has been used in numerous past studies of coccidioidomycosis. This system comprises the sum of points assigned based on the findings of: (1) clinical assessments, (2) radiographic imaging, and (3) serologic assays, with a lower score indicating better health.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events | 180 days
  Treatment-emergent adverse events are defined as new events that occur following subject entry into the study or events that worsen following study entry state. Severity grading will be based on Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. This is a descriptive scoring system which can be used for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term as follows: Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE; Grade 5 = Death related to AE.
Number of Participants with Abnormal Laboratory Evaluations of Safety | 180 days
  Abnormal is defined as at least a 1 grade shift from baseline. Severity grading will be based on Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. This is a descriptive scoring system which can be used for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term as follows: Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE; Grade 5 = Death related to AE.
Number of Participant Discontinuations of Therapy Due to Treatment-Emergent Adverse Events and/or Laboratory Evaluations of Safety | 180 days
  Number of Participant Discontinuations of Therapy Due to Treatment-Emergent Adverse Events and/or Laboratory Evaluations of Safety
Number of Participants with Any Interruptions of Therapy due to Treatment-Emergent Adverse Events and/or Abnormal Laboratory Evaluations of Safety | 180 days
  Number of Participants with Any Interruptions of Therapy due to Treatment-Emergent Adverse Events and/or Abnormal Laboratory Evaluations of Safety
Number of Participants with Interruptions of Therapy 7 Days or More in Duration due to Treatment-Emergent Adverse Events and/or Abnormal Laboratory Evaluations of Safety | 180 days
  Number of Participants with Interruptions of Therapy 7 Days or More in Duration due to Treatment-Emergent Adverse Events and/or Abnormal Laboratory Evaluations of Safety
Mean, Median, and Quartile Score Values for Mental Component Summary and Physical Component Summary Scores of the SF-12v2 Survey | 42 days
  The Short Form 12 Question Health Survey, version 2 (SF-12v2) is a 12-question multipurpose survey instrument derived from the larger, Short Form 36 Question Survey. The SF-12v2 is to help determine the participant's overall state of wellbeing and health-related quality of life by means of assessing both physical and mental status at the time of the survey. The 8 domains of the survey are: physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role- emotional (RE), and mental health (MH). Mental and physical composite scores (MCS & PCS) are computed using the scores of twelve questions. MCS and PCS values can range from 0 to 100, where a higher score indicates better health.
Mean, Median, and Quartile Score Values for Mental Component Summary and Physical Component Summary Scores of the SF-12v2 Survey | 180 days
  The Short Form 12 Question Health Survey, version 2 (SF-12v2) is a 12-question multipurpose survey instrument derived from the larger, Short Form 36 Question Survey. The SF-12v2 is to help determine the participant's overall state of wellbeing and health-related quality of life by means of assessing both physical and mental status at the time of the survey. The 8 domains of the survey are: physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role- emotional (RE), and mental health (MH). Mental and physical composite scores (MCS & PCS) are computed using the scores of twelve questions. MCS and PCS values can range from 0 to 100, where a higher score indicates better health.

CONTACTS AND LOCATIONS:
Overall Officials: George R Thompson, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No